CLINICAL TRIAL: NCT01114009
Title: Effects of Recruitment Maneuvers in Early ALI and ARDS Patients
Brief Title: Effects of Recruitment Maneuvers in Early Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LUN WEI LIU (Other)
Collaborators: Chi Mei Medical Hospital (Other)
Responsible Party: Sponsor-Investigator, LUN WEI LIU, Chi Mei Medical Hospital, Chi Mei Medical Hospital
Organization: Chi Mei Medical Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLFHR9803
Record Dates: First submitted 2010-04-26; First posted 2010-04-30 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Acute Respiratory Distress Syndrome; Lung Injury, Acute
Keywords: recruitment maneuvers; ARDS; lung protective strategy; ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lung recruitment maneuver (Experimental): The maneuver briefly increases the alveolar pressure to open recruitable lung (50 cmH2O), sustained with adequate positive end-expiratory pressure(PEEP) after lung recruitment, to avoid derecruitment.
  Interventions: Procedure: Lung recruitment maneuver; Procedure: Lung protective strategy group
- Lung protective strategy (Active Comparator): Lung protective strategy group received lung protective strategy without recruitment maneuver
  Interventions: Procedure: Lung protective strategy group

INTERVENTIONS:
Procedure: Lung recruitment maneuver — Lung recruitment maneuver conducted with a PEEP 35 cmH2O and peak inspiration pressure up to 50 cmH2O maintain 2 mins, then find the closing pressure (if possible), after that, PEEP is set higher 2 cmH2O above closing pressure
  Arms: Lung recruitment maneuver
Procedure: Lung protective strategy group — Lung protective strategy group received Lung protective strategy without recruitment maneuver

SUMMARY:
The purpose of this study is to evaluate the effect of lung recruitment maneuver in patients with early ALI/ARDS

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) was first described in the medical literature in 1967. Patients with ARDS mostly require mechanical ventilatory support due to hypoxic respiratory failure. Mechanical ventilation can induce lung injury (ventilator-induced lung injury, VILI) by causing overdistention and repetitive opening and closing of unstable lung units. Data from a number of randomized controlled trials indicate that a lung protective ventilatory strategy with small tidal volume and low plateau pressure reduces mortality in acute lung injury (ALI) and acute respiratory distress syndrome. Lung recruitment maneuvers are being used in the management of ALI and ARDS, but recruitment maneuvers are still controversial. Lung recruitment maneuver is aimed to open the collapsed lung and keep the lung open. The maneuver briefly increases the alveolar pressure to open recruitable lung, sustained with adequate positive end-expiratory pressure(PEEP) after lung recruitment, to avoid derecruitment. We want to enroll 120 patients with early ALI/ARDS in this randomized controlled study. The study group use recruitment maneuver and lung protective ventilatory strategy, and the control group use lung protective ventilatory strategy only. Concerning about both safety and efficacy, we design a modified recruitment maneuver protocol which has never been published in previous medical literature. The primary outcome is ventilator-free days and ICU-free days, and secondary outcomes include ventilator weaning rate, and 28-day mortality and cost effectiveness analysis. Since no randomized controlled trials clearly establish benefit from recruitment maneuvers, we hope this study would be able to provide some evidence on whether lung recruitment should be used in the routine management of ALI/ARDS.

ELIGIBILITY:
Inclusion Criteria:

* met criteria of ALI/ARDS
* PaO2/FiO2 less than or equal 250 mmHg after standard ventilator setting (FiO2 more than or equal 0.5 and PEEP more than or equal 10 cmH2O)at least 30 mins

Exclusion Criteria:

* age less than 18 years
* duration of mechanical ventilator more than 72 hours
* Pneumothorax or subcutaneous emphysema or bullous lung disease
* severe chronic respiratory disease
* intracranial hypertension or received craniotomy surgery
* longterm dependent ventilator
* Neuromuscular disease
* premorbid conditions with an expected 6 month mortality risk exceeding 50%

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
28-day hospital mortality | Two year

SECONDARY OUTCOMES:
Ventilator-free days | Two year
Ventilator weaning rate | Two years
Cost-effectiveness analysis | Two years
ICU-free days | Two years

CONTACTS AND LOCATIONS:
Overall Officials: WEI LUN LIU, MD, Principal Investigator — Chi Mei Medical Center, Liou Ying
Locations (1):
- Chi Mei Medical Center,Liou Ying, Tainan, Taiwan